CLINICAL TRIAL: NCT03142789
Title: Comparison of the Analgesic Effect of an ACB (Adductor Canal Block) Using a New Suture-method Catheter vs a Standard Perineural Catheter vs a Single Bolus: A Randomized, Blinded, Controlled Study
Brief Title: Adductor Canal Block After Total Knee Replacement - a Suture-method Catheter vs a Standard Catheter vs a Single Bolus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Ulrik Grevstad, MD, phd, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EudraCT number: 2016-005069-30
Record Dates: First submitted 2017-05-01; First posted 2017-05-05 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Pain Management
Keywords: Pain; Total knee arthroplasty; Regional anesthesia
MeSH Terms: conditions — Agnosia; Pain | interventions — cerivastatin

STUDY DESIGN:
Intervention Model Description: The study is performed as a blinded, randomized, controlled study. Randomization will be based on a computer-generated block randomization list in a 1:1:1 ratio, block sizes of 9. A person, not otherwise involved in the study, will prepare the randomization list and keep it, locked away in a secure place. 2 sets of consecutively numbered, sealed, opaque, code envelopes will be prepared by the same person.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Please see "Model Description"
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Certa Catheter (Active Comparator): A Certa-catheter (suture method) is inserted under ultrasound guidance at the midthigh level in the adductor canal, using an in plane technique, short/oblique axis view.
  A bolus of ropivacaine will be administered during real time US imaging to ensure correct placement of the catheter (initial bolus). An infusion pump will be connected immediately following catheter insertion, delivering intermittent boluses every 8 hours until 12 pm on POD2.
  2 dressings will be applied (medial and lateral) to obscure which catheter has been placed.
  Interventions: Drug: Initial bolus (Certa and standard catheter groups); Drug: Intermittent boluses (Certa and standard catheter groups)
- Standard Catheter (Active Comparator): A Standard-catheter is inserted under ultrasound guidance at the midthigh level in the adductor canal, using an in plane technique, short/oblique axis view.
  A bolus of ropivacaine will be administered during real time US imaging to ensure correct placement of the catheter (initial bolus). An infusion pump will be connected immediately following catheter insertion, delivering intermittent boluses every 8 hours until 12 pm on POD2.
  2 dressings will be applied (medial and lateral) to obscure which catheter has been placed.
  Interventions: Drug: Initial bolus (Certa and standard catheter groups); Drug: Intermittent boluses (Certa and standard catheter groups)
- Single Bolus (Active Comparator): A bolus of ropivacaine will be injected into the adductor canal, at the midthigh level, using a 80 mm x 22G Pajunk needle during real time US imaging (initial bolus).
  A sham catheter (25 Certa and 25 standard catheters according to randomi-zation) will be fixed externally and covered by dressings as in the catheter groups groups (Certa and standard). Care will be taken to use approximately the same amount of time as used in the catheter groups (Certa and standard) An infusion pump will be connected immediately following catheter insertion, delivering intermittent boluses into the dressing every 8 hour until 12 PM on POD2.
  Interventions: Drug: Initial bolus (Single bolus group); Drug: Intermittent boluses (Single bolus group)

INTERVENTIONS:
Drug: Initial bolus (Certa and standard catheter groups) — 10 ml of ropivacaine 0,75% will be used to ensure correct position of the needle and to expand the adductor canal, followed by injection of another 10 ml of ropivacaine 0.75% via the catheter during real time US imaging to ensure correct placement of the catheter.
  Arms: Certa Catheter; Standard Catheter
Drug: Initial bolus (Single bolus group) — 20 ml of ropivacaine 0.75%
  Arms: Single Bolus
Drug: Intermittent boluses (Certa and standard catheter groups) — 20 ml of ropivacaine 0.2% every 8 hour in the catheter
  Arms: Certa Catheter; Standard Catheter
Drug: Intermittent boluses (Single bolus group) — 0.1ml of ropivacaine 0.2% every 8 hour in the sham catheter
  Arms: Single Bolus

SUMMARY:
In this study we wish to investigate the analgesic effect of the administration of 0.2% ropivacaine for an adductor canal block as repeated boluses (20 ml every 8 hours) through a new suture-method catheter or a standard perineural catheter compared with a single bolus (20 ml), in patients following primary total knee arthroplasty.

DETAILED DESCRIPTION:
The aim of the study is to compare the clinical effects of three different administration forms for an ACB: repeated intermittent boluses through a Certa catheter (CC) versus repeated boluses through a standard catheter (through the needle) (SC) versus a single bolus (SB). Our dual hypothesis is that repeated boluses through a catheter (either Certa or standard catheter) reduces opioid consumption (primary outcome), as well as reduces pain scores, enhances ambulation and muscle strength compared with a single bolus, and that the Certa catheter is superior to a standard catheter.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for unilateral total knee arthroplasty in spinal anesthesia
* Patients who gave their written informed consent to participating in the study after having fully understood the contents of the protocol and restrictions
* ASA 1-3
* Ability to perform a TUG test preoperatively

Exclusion Criteria:

* Patients who cannot cooperate
* Patients who cannot understand or speak Danish.
* Patients with allergy to the medicines used in the study
* Patients with a daily intake of strong opioids (morphine, oxycodone, ketobemidone, methadone, fentanyl) during the last 4 weeks
* Patients suffering from alcohol and/or drug abuse - based on the investigator's assessment
* Rheumatoid arthritis
* BMI > 40
* Neuromuscular pathology in the lower limbs
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | from end of surgery until 12 (noon) on POD 2 (Postoperative Day)
  • Total opioid consumption (PCA pump and any potential rescue administration) between groups (SB vs CC, SB vs SC and CC vs SC)

SECONDARY OUTCOMES:
VAS (Visual analog scale) flexion | o Pain is recorded preoperatively before administration of medication, and postoperatively at the PACU (Postoperative Care Unit), at 8 PM on the day of surgery, at 8 AM, 12 (noon) and 8 PM on POD 1 and finally at 8 AM and 12 (noon) on POD 2.
  VAS pain score (0-100mm) during 45 degrees active knee flexion
VAS rest | o Pain is recorded preoperatively before administration of medication, and postoperatively at the PACU, at 8 PM on the day of surgery, at 8 AM, 12 (noon) and 8 PM on POD 1 and finally at 8 AM and 12 (noon) on POD 2.
  VAS pain score (0-100mm) during rest
VAS-TUG (Time-Up-and-Go-Test) | 12 (noon) on POD 1 and 2
  Worst VAS pain score (0-100mm) during Timed-Up-and-Go test
TUG-test | 12 (noon) on POD 1 and 2
  Timed-Up-and-Go test
6 minutes walk test | 12 (noon) on POD 1 and 2
  How many meters the patient can walk (using a high 4-wheel walker) in 6 minutes
MVIC (Maximum Voluntary Isometric Contraction) | Preoperatively and at 12 (noon) on POD 1 and 2
  Quadriceps strength assessed as maximum voluntary isometric contraction in percentage of preoperative baseline values.
TUG test, patient number | 12 (noon) on POD 1 and 2
  Number of patients able to perform the TUG test using a high 4-wheel walker

OTHER OUTCOMES:
Catheter testing - temperature | preoperatively and at 12 (noon) on POD 1 and 2
  Using an alcohol swab we will test for temperature discrimination ability in the saphenous distribution area
Catheter testing - Ultrasound | on POD 2 at 2 PM
  At the end of the study period all patients will have an US evaluation of the catheters (a sham evaluation in the SB group) by one of the unblinded investigators. 20 ml of ropivacaine 0.2% will be injected during real-time US visualization. Spread outside the canal will be noted. In case the patient has a displaced catheter repositioning will be attempted, whether repositioning is possible is noted on a separate CRF (Case Report Form). The following will be noted; is the orifice of the catheter visible (yes/no), does injection result in a spread in-side the adductor canal (yes/no), can the catheter be repositioned to obtain a spread inside the canal (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Grevstad, MD, phd, Principal Investigator — Gentofte Hospital
Locations (1):
- Gentofte Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
We have not yet decided whether IPD will be made available to other researchers

REFERENCES:
- [Derived] Lyngeraa TS, Jaeger P, Gottschau B, Graungaard B, Rossen-Jorgensen AM, Toftegaard I, Grevstad U. Comparison of the analgesic effect of an adductor canal block using a new suture-method catheter vs. standard perineural catheter vs. single-injection: a randomised, blinded, controlled study. Anaesthesia. 2019 Nov;74(11):1397-1405. doi: 10.1111/anae.14814. Epub 2019 Aug 29. PMID 31465115